CLINICAL TRIAL: NCT03558412
Title: A Clinical Trial of Decitabine Combined With CODOX-M/IVAC in Relapsed or Refractory T-lymphoblastic Lymphoma
Brief Title: A Clinical Trial of Decitabine in Relapsed or Refractory T-lymphoblastic Lymphoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mingzhi Zhang (Other)
Responsible Party: Sponsor-Investigator, Mingzhi Zhang, The director of oncology department of the first affiliated hospital, Zhengzhou University
Organization: Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hnslblzlzx20171118
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: T-lymphoblastic Lymphoma
Keywords: Decitabine; RR; TTP; OS; MST
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Arm A (Experimental): Decitabine+CODOX-M/IVAC for patients with relapsed or refractory T-lymphoblastic lymphoma who used Hyper-CVAD or BFM-90 as first-line therapy:regimen A:CODOX-M:cyclophosphamide,epirubicin,vincristine,methotrexate.Regimen B :IVAC:ifosfamide,etoposide，cytarabine.Decitabine,10mg,ivgtt,used for 5 days before A+B.
  Interventions: Combination Product: CODOX-M/IVAC; Drug: Decitabine

INTERVENTIONS:
Combination Product: CODOX-M/IVAC — Given ivgtt
Drug: Decitabine — Given ivgtt
  Other Names: 5-Aza-2'-deoxycytidine

SUMMARY:
To explore the safety, tolerability, and clinical effects of decitabine combined with Second-line chemotherapy regimens for patients with relapsed or refractory T-lymphoblastic lymphoma.

DETAILED DESCRIPTION:
This is a prospective, open，investigator initial clinical trial with a single arm, aimed to evaluate the safety, tolerability, and efficacy of decitabine combined with Second-line chemotherapy regimens (CODOX-M/IVAC) in relapsed or refractory T-lymphoblastic lymphoma. A total of 40 patients are planned to be enrolled into the study. Patients with diagnosis of relapsed or refractory T-lymphoblastic lymphoma will be treated with decitabine plus CODOX-M/IVAC. The primary end point is responder rate (RR) and time to progression (TTP), and the secondary end points include overall survival (OS) and the median survival time (MST).

ELIGIBILITY:
Inclusion Criteria:

* age: 14~60 years; ECOG rate ≤ 2; expected survival > 3 months;
* patients with T-lymphoblastic lymphoma diagnosed by histopathology detection;
* patients ever received chemotherapy and/or radiotherapy;and can not be transplanted hematopoietic stem cells;
* patients with no chemotherapy contraindications: hemoglobin ≥ 90 g/L, absolute neutrophil count ≥1.5 x 109/L, blood platelet ≥100 x 109/L, ALT and AST ≤ 2-fold upper normal limit, serum bilirubin ≤ 1.5-fold upper normal limit, serum creatinine ≤ 1.5-fold upper normal limit, serum albumin ≥ 30 g/L, normal serofibrinogen;
* at least one measurable nidus;
* no other severe diseases conflict with this project, cardiopulmonary function is basically normal;
* the urine or blood pregnancy test of women in childbearing age must be negative in 7 days before follow-up visit;
* applicable for follow-up visit;
* no other antitumor adjoint therapy (including antitumor Chinese medicine, immunotherapy and biotherapy), but double phosphate anti-bone transfer therapy and other symptomatic treatment are acceptable;
* understanding this study and assigning informed consent.

Exclusion Criteria:

* rejecting providing blood preparation;
* allergic to drug in this study and with metabolic block;
* rejecting adopting reliable contraceptive method in pregnancy or lactation period;
* uncontrolled internal medicine disease (including uncontrolled diabetes, severe incompetence cardiac, lung, liver and pancreas);
* with severe infection;
* with primary or secondary central nervous system tumor invasion;
* with immunotherapy or radiotherapy contraindication;
* ever suffered with malignant tumor;
* having peripheral nervous system disorder or dysphrenia;
* with no legal capacity, medical or ethical reasons affecting research proceeding;
* participating other clinical trials simultaneously;
* adopting other anti-tumor medicine excluding this research;
* the researchers considering it inappropriate to participate in the study.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
RR | up to 2 months
  Responder Rate
TTP | up to 2 months
  Time To Progression

SECONDARY OUTCOMES:
OS | up to 2 months
  Overall Survival
MST | up to 2 months
  Median Survival Time

CONTACTS AND LOCATIONS:
Overall Officials: Mingzhi zhang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Oncology Department of The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China